CLINICAL TRIAL: NCT01939054
Title: A Randomized, Controlled, Open-Label, Multicenter, Phase 2 Study of Nimotuzumab Plus Docetaxel and Capecitabine Versus Docetaxel and Capecitabine as First-Line Treatment in Patients With Recurrent/Metastatic Triple Negative Breast Cancer
Brief Title: Nimotuzumab Plus Docetaxel and Capecitabine Versus Docetaxel and Capecitabine in the Treatment of Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Principal Investigator, Binghe Xu, Director of Medical Oncology, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-BC-001
Record Dates: First submitted 2013-08-28; First posted 2013-09-11 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — nimotuzumab; Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nimotuzumab,docetaxel,capecitabine (Experimental): Nimotuzumab 400mg/w,IV,once a week and Docetaxel 75 mg/m2,IV,D1, every 21 days a cycle and Capecitabine 1000mg/m2, orally, twice daily, D1-D14
  Interventions: Drug: Nimotuzumab; Drug: docetaxel; Drug: capecitabine
- docetaxel,capecitabine (Active Comparator): Docetaxel 75 mg/m2,IV,D1, every 21 days a cycle and Capecitabine 1000mg/m2, orally, twice daily, D1-D14
  Interventions: Drug: docetaxel; Drug: capecitabine

INTERVENTIONS:
Drug: Nimotuzumab
  Arms: Nimotuzumab,docetaxel,capecitabine
Drug: docetaxel
Drug: capecitabine

SUMMARY:
Nimotuzumab is an IgG1 humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR), inhibiting tyrosine kinase activation. This is a randomized, controlled, open-Label, multicenter, phase Ⅱ clinical trial of nimotuzumab plus Docetaxel and Capecitabine（TX）versus Docetaxel and Capecitabine（TX）as first-line treatment in patients with recurrent/metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
The control group received docetaxel + capecitabine regimen;Experimental group received Nimotuzumab combined docetaxel + capecitabine regimen.The main purpose is to evaluate Nimotuzumab Plus Docetaxel and Capecitabine（TX）as First-Line Treatment in Patients With Recurrent/Metastatic triple negative breast cancer would improve objective response rate (ORR ) comparing with Docetaxel and Capecitabine（TX）.

ELIGIBILITY:
Inclusion Criteria:

1. Histological and immunohistochemistry (IHC) confirmed recurrent or metastatic triple-negative breast cancer .
2. Previous chemotherapy should include anthracycline or taxane; No prior chemotherapy after metastasis.
3. Females with age between 18 and 70 years old
4. ECOG performance status 0 or 1.
5. At least one measurable disease according to the response evaluation criteria in solid tumor (RECIST) by magnetic resonance imaging, or computed tomography; The target lesions is Unresectable; The target lesions did not receive radiotherapy or relapse within the radiation field;
6. Life expectancy ≥ 12 weeks.；
7. WBC count ≥ 4 × 109 / L, neutrophils ≥ 1.5 × 109 / L, platelet count ≥ 100 × 109 / L, hemoglobin ≥ 6.21mmol / L (10 g / dL);
8. Total bilirubin (TBL)≤ 1.5 x ULN (upper limit of normal reference values); AST and ALT ≤ 2.5 x ULN or ≤ 5 ULN (Liver metastasis);Serum creatinine ≤ 1.5 x ULN.
9. Before enrollment, patients have fully recovered from previous treatment-related toxicity;
10. Subjects with fertility must accept effective contraceptive measures;
11. Signed informed consent

Exclusion Criteria:

1. Previously treatment regimen including anti EGFR monoclonal antibody;
2. Receiving other anti-cancer medicine treatment during the study
3. Participate in other clinical trials within 4 weeks in this group;
4. Accepted taxane treatment in 1 year;
5. Presence of neurological symptoms due to brain metastasis, patients receiving steroidal anti-edema drugs therapy;
6. Patients having a history of clinically significant symptomatic angina, arrhythmia or congestive heart failure without control;
7. Diagnosed with severe interstitial pneumonitis or pulmonary fibrosis by chest CT;
8. Pleural effusion, ascites require to be drained;
9. Adverse drug addiction and drug abuse, long-term alcoholics, as well as AIDS patients; patients with severe or uncontrolled complications, such as infection requiring systemic therapy, fever (≥ 38 ℃), diabetes or hypertension can not be controlled by medicine, other complications may interfere with drug therapy;
10. Patients with a history of drug allergy (≥ CTCAE 2 level) such as shock or allergic symptoms, especially have allergic reactions to similar drugs in the past, have severe allergies reactions to drugs containing polysorbate eighty (Tween 80);
11. Uncontrolled seizures or loss of insight due to mental disorders;
12. Pregnant or lactating women；
13. Researchers think improper for this trial

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
ORR | every six weeks, up to 1 year
  Evaluation ORR every six weeks,with RECIST 1.1.

SECONDARY OUTCOMES:
PFS | every six weeks, up to 1 year
Number and ratio of AEs | up to 1 year
  Observe and record AEs when AEs occurred
Relationship of tissue/serum EGFR between efficacy and prognosis | 1 year
  every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Principal Investigator — Cancer Insititute and Hospital, CAMS
Locations (9):
- China (9):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing cancer hospital, Beijing, Beijing Municipality
  - The General Hospital of the People's Liberation Army (PLAGH), Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - FuDan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Xijing Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of College of Medicine, Zhejiang University (First Hospital of Zhejiang Province), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang